CLINICAL TRIAL: NCT05710965
Title: A Randomized Controlled Intervention Study to Assess a Wearable Digital Therapy for Youth With ADHD
Brief Title: Assessing a Wearable Digital Therapy for Youth With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revibe Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RV-003
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FRx-001 (Active Comparator): FRx-001 is a wearable digital intervention that provides therapeutic vibrations to the subjects wrist and scheduled assistive messaging.
  Interventions: Device: FRx-001
- FRx-003 (Active Comparator): FRx-003 is a wearable digital intervention that provides therapeutic vibrations to the subjects wrist and may include periodic assistive messaging.
  Interventions: Device: FRx-003
- FRx-004 (Active Comparator): FRx-004 is a wearable digital intervention that displays periodic therapeutic assistive messaging.
  Interventions: Device: FRx-004

INTERVENTIONS:
Device: FRx-001 — Wearable digital therapy
  Arms: FRx-001
Device: FRx-003 — Wearable digital therapy
  Arms: FRx-003
Device: FRx-004 — Wearable digital therapy
  Arms: FRx-004

SUMMARY:
The purpose of this study is to evaluate and compare three different investigational wearable digital interventions to determine if they are helpful for improving symptoms and functioning in children diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
The study is a randomized controlled trial of three investigational wearable digital therapies. An online screening questionnaire will evaluate eligibility for the study. Parents and teachers will complete baseline measures, after which the child will wear the assigned device to school Monday-Friday for a four-week period. Parents and teachers will complete the measures again at the end of the four-week intervention period. Compliance with wearing the device will be monitored remotely.

ELIGIBILITY:
Inclusion Criteria:

Youth Participants

* Parent-reported diagnosis of ADHD
* Must be between the ages of 8 and 12 years of age
* Must live in the United States
* Must be able to understand English well
* Must be able to read English well (reading at grade level independently or with adult assistance)
* Must be attending in-class (as opposed to hybrid or virtual) school during the period of the trial
* Must be willing to wear the device to school on their wrist Monday to Friday for a period of four-weeks
* Parent-rated ADHD-RS-5 Total score of ≥ 28*

  * The ADHD-RS-5 score will be determined based on the ratings provided in the parent baseline questionnaire. Any youth with a parent-rated Total score <28 will be allowed to remain in the study but will not be included in the per protocol analyses.

Parent Participants

* Must be 18 years of age or older
* Must be willing to invite the child's teacher to participate
* Must live in the United States
* Must read and understand English well
* Must have a mobile device that can be used to download and install the software application and sync to the device
* Must be willing to have their child wear the device to school Monday to Friday for a period of four weeks and sync and charge the device

Teacher Participants

* Must be 18 years of age or older
* Must live in the United States
* Must have known the student for at least four weeks
* Must read and understand English well
* Must be providing in person classroom learning to the youth during the study period

Exclusion Criteria:

Youth Participants

* Motor condition (e.g., physical deformity of the hands/arms; prostheses) that prevents tapping the device if prompted or unable to feel vibrations from the device on their wrist (should there be any), as reported by the parent.
* Home schooled
* Diagnosed (parent-reported) Autism Spectrum Disorder, Intellectual Disability, Pervasive Developmental Disorder, Schizophrenia Spectrum Disorder.
* Not undergoing pharmacological treatment for ADHD (currently or in the past 30 days)
* Has ever worn or used Revibe Connect prior to the study or has a sibling who has
* Has ever participated in a research study conducted by Revibe Technologies or has a sibling who has
* Has a sibling participating in the study. Only one child per family is eligible to participate.
* Allergy to latex (parent-reported)

Parent and Teacher Participants

• No exclusion criteria other than not meeting the inclusion criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale-5 (ADHD-RS-5), School Version: Inattention Subscale | Change from Baseline to Post-intervention (4 weeks)
  Nine teacher rated items aligned with Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) Inattentive symptoms, scored on a 4-point Likert scale from "never or rarely" to "very often". Scores range from 0-27, higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
ADHD Rating Scale-5, Home Version: Inattention Subscale | Change from Baseline to Post-intervention (4 weeks)
  Nine parent rated items aligned with DSM-5 Inattentive symptoms, scored on a 4-point Likert scale from "never or rarely" to "very often". Scores range from 0-27, higher scores indicate greater symptom severity.
ADHD Rating Scale-5, School Version: Total score | Change from Baseline to Post-intervention (4 weeks)
  Sum of the teacher rated Inattentive and Hyperactivity-Impulsivity Subscale scores. Scores range from 0-54, higher scores indicate greater symptom severity.
ADHD Rating Scale-5, Home Version: Total score | Change from Baseline to Post-intervention (4 weeks)
  Sum of the parent rated Inattentive and Hyperactivity-Impulsivity Subscale scores. Scores range from 0-54, higher scores indicate greater symptom severity.

OTHER OUTCOMES:
ADHD Rating Scale-5, School Version: Hyperactivity-Impulsivity Subscale | Change from Baseline to Post-intervention (4 weeks)
  Nine teacher rated items aligned with DSM-5 Hyperactivity-Impulsivity symptoms, scored on a 4-point Likert scale. Scores range from 0-27, higher scores indicate greater symptom severity.
ADHD Rating Scale-5, Home Version: Hyperactivity-Impulsivity Subscale | Change from Baseline to Post-intervention (4 weeks)
  Nine parent rated items aligned with DSM-5 Hyperactivity-Impulsivity symptoms, scored on a 4-point Likert scale. Scores range from 0-27, higher scores indicate greater symptom severity.
Conners 4, Short Form: Parent | Change from Baseline to Post-intervention (4 weeks)
  Parent completed ratings of ADHD symptoms and functioning. Items are rated on a 4-point Likert scale. Subscale raw scores are converted to T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate greater symptom severity or impairment.
Conners 4, Short Form: Teacher | Change from Baseline to Post-intervention (4 weeks)
  Teacher completed ratings of ADHD symptoms and functioning. Items are rated on a 4-point Likert scale. Subscale raw scores are converted to T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate greater symptom severity or impairment.
Comprehensive Executive Function Inventory: Parent | Change from Baseline to Post-intervention (4 weeks)
  Parent completed ratings of a child's executive function. Consists of 9 domains and a total score. Items are rated on a 6-point Likert scale. Subscale raw scores are converted to standard scores with a mean of 100 and standard deviation of 15. Higher scores are indicative of better functioning.
Comprehensive Executive Function Inventory: Teacher | Change from Baseline to Post-intervention (4 weeks)
  Teacher completed ratings of a child's executive function. Consists of 9 domains and a total score. Items are rated on a 6-point Likert scale. Subscale raw scores are converted to standard scores with a mean of 100 and standard deviation of 15. Higher scores are indicative of better functioning.
Impairment Rating Scale - Parent | Change from Baseline to Post-intervention (4 weeks)
  Parent completed ratings of impairment in youth with ADHD. Parent version includes 8 items. The 8th represents overall impairment. Ratings are made on a 7-point Likert scale from "no problem/definitely does not need treatment or special services" to "extreme problem/definitely needs treatment or special services". Higher scores indicate more severe problems.
Impairment Rating Scale - Teacher | Change from Baseline to Post-intervention (4 weeks)
  Teacher completed ratings of impairment in youth with ADHD. Teacher version includes 7 items. The 7th represents overall impairment. Ratings are made on a 7-point Likert scale from "no problem/definitely does not need treatment or special services" to "extreme problem/definitely needs treatment or special services". Higher scores indicate more severe problems.
Weiss Functional Impairment Rating Scale - Parent Form | Change from Baseline to Post-intervention (4 weeks)
  Parent completed ratings of child's overall functioning across six domains including a total score. Items are rated on a 4-point Likert scale ranging from "not at all or never" to "very much or very often", as well as a "not applicable" option. Higher scores are associated with impairment.
Academic Performance Rating Scale | Change from Baseline to Post-intervention (4 weeks)
  A 19-items scale developed to reflect teachers' perceptions of children'ts academic performance and abilities in classroom settings. Items are rated on a 5-point Likert scale, and scores are summed for each of the factor scores: Academic Success, Impulse Control, and Academic Productivity. A total score is also calculated for overall academic performance. Higher scores are representative of stronger classroom functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Revibe Technologies, Wake Forest, North Carolina, United States